CLINICAL TRIAL: NCT04092296
Title: Efficacy of Resin Infiltration of Proximal Caries Tested With DIAGNOcam and Bitewing Radiography:Randomized Controlled Clinical Trial
Brief Title: Efficacy of Resin Infiltration of Proximal Caries
Acronym: RIDCBW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Fei Wang, graduate student, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20180103
Record Dates: First submitted 2019-09-14; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Caries; Initial
MeSH Terms: interventions — Tooth Remineralization; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resin infiltration (Experimental): resin infiltrant (Icon product, DMG, Hamburg,Germany)
  Interventions: Other: resin infiltration
- remineralization (Active Comparator)
  Interventions: Other: remineralization; Other: sham

INTERVENTIONS:
Other: resin infiltration — using infiltrant resin intervene proximal caries
  Arms: resin infiltration
Other: remineralization — using fluoride to remineralize proximal caries
  Arms: remineralization
Other: sham — replace resin with water
  Arms: remineralization

SUMMARY:
The aim of the present study was to assess the clinical efficacy of resin infiltration of interproximal caries lesions using a novel measure method-----DIAGNOcam. This study is conducted on adults (15-40y）with the aim of comparing the therapeutic effects of infiltrating caries lesions and fluoride remineralization treatment after 1, 2, and 3 yrs. The outcome (lesion progression) is evaluated by DIAGNOcam and radiographic techniques.And we would compare the sensitivity of monitoring progression of caries between DIAGNOcam and bitewing radiography.

DETAILED DESCRIPTION:
On the baseline,At a screening visit, eligibility of interested participants is checked with DIAGNOcam by a researcher(WF),in addition,a pair of standardized conventional bitewing radiographs is taken using a film holder Kwik-Bite by a very experienced dental assistant .

two reviewers(SC、XYJ) who are trained the scoring systems score the DIAGNOcam and bitewing image independently,disagreements are solved by consensus and a final DIAGNOcam and bitewing score are given.Participants who have two E2 lesions are picked to join the first set up.

A.DIAGNOcam image scoring system:

E1:Dark shadow confined to the out half of the enamel E2:Dark shadow confined to the inner half of the enamel D1:Dark shadow reach dentin ,dentin caries penetrating the enamel-dentin junction linerly D2:Deep dentin are involved

B .bitewing radiograph scoring system:

E1 = radiolucency in the out half of the enamel; E2 = radiolucency extending to the enamel dentine junction; D1= radiolucency into dentine but limited to the outer third; D2 = radiolucency into middle or middle third of the dentine; D3 = radiolucency into middle or inner third of the dentine; 2.3 Caries risk and periodontal condition assessment On the baseline ,we use the dmft/s to asess the caries risk.In addition,Occurrence of plaque is scored as 0 = no visible plaque or 1 = visible plaque; the status of the gingiva is scored as 0 = sound, 1 = redness, with no bleeding after probing, 2 = bleeding after probing, and 3 = heavily inflamed.

2.4 Allocation From each pair, 1 lesion is allocated to the "test" and 1 to the "control" group using random number table and sealed in opaque envelope to prevent the allocation being known in advance of, or during, enrolment 2.5 Treatment INTERVENTION 1:Resin infiltration:Treatment is performed by a single trained investigator (WF) at the Wuhan University stomatological Hospital . A rubber dam is applied to achieve dry working conditions. In the test group, allocated teeth are slightly separated by plastic wedges (Wedge Wands, small or medium; Garrison, Übach-Palenberg, Germany) that have been flattened by a scalpel to leave space below the contact point. A piece of polyurethane foil is placed in the contact area with a plastic holder to protect the adjacent tooth. A 15% HCl etching gel (Icon product, DMG, Hamburg,Germany) is applied by syringe in the area below the contact point for 120 sec. Subsequently, the gel is washed off with air-water-spray for 30 sec. The lesion is desiccated by air-blowing for 30 sec, application of ethanol for 30 sec, and air- blow ing again for 30 sec. An infiltrant (Icon product,DMG) is applied with another plastic holder,in this time the investigator need to shut off the light.. After 3 min of penetration time, excess material is removed by air blowing and flossing, and the resin is light-cured for 1 min from the buccal, occlusal, and oral aspects. The infiltration step is repeated once with a penetration time of 1 min to infiltrate remaining porosities.

To avoid behavioral changes of participants with regard to oral hygiene, we will not inform them about the treatment allocation of their teeth. To ensure blinding, we perform a placebo treatment on control teeth: Instead of HCl-gel and infiltrant, water is used. Fluoridation, oral hygiene, and dietary instructions are given to the patients.

After the application of the infiltrant,and restoration,we will check with DIAGNOcam and Bitewing radiography again,because we have no idea about the characteristics of the DIAGNOcam image after resin infiltration.

2.6 Follow-up Examination Every three months since then, participants will be re-called for follow-up examination. DIAGNOcam and bitewing examinations are operated by the same investigator(WF) and the same experienced dental assistant .

Clinical examination and caries risk assessment are performed by one clinical investigator (YCC), who is blinded with regard to treatment group allocation of teeth.

The primary outcome is the progression of lesion depth, assessed by pair-wise comparison DIAGNOcam and pair-wise comparison of the bitewing radiographs .

Secondary outcome

1. Patients will be interviewed for possible unwanted side-effects.
2. Participant and operator perception, as measured by standardised/validated questionnaires
3. The sensitivity of DIAGNOcam and bitewing radiography in monitoring caries' progression.

Additional follow-up examinations are planned 24 and 36 months after intervention.

If a lesion of any group progresses during the follow-up period radiographically to the D2 or D3 stage, restorative treatment will be performed.

In order to allow for reproducible DIAGNOcam geometry, the handled camera keeps vertical to the tooth long axis.

DIAGNOcam images as well as bitewing radiographs will be assessed by two reviewers(SC,XYJ) independently (inter-examiner reliability was assessed), both of whom are blinded with regard to treatment group allocation. Both assessors attend a training and calibration session one day prior to examination. By anonymising the radiographs, masking the stage of treatment (i.e. baseline or follow-up) or both to ensure adequate blinding of assessors.First, the DIAGNOcam and radiographic stage (E1-D3) of lesions at baseline and follow-up examination was assessed. Subsequently, examiners read the DIAGNOcam images and radiographs pairwise and judged whether lesions showed progression, regression, or were stable. In cases of different interpretation between examiners, a consensus rank was agreed. To assess intra-observer reliability, we repeated the readings after 4 wks.

3.Statistical Analysis Inter- as well as intra-observer reliability was assessed by kappa statistics. We used the X2test to analyze differences between treatment and control groups with regard to lesion progression (pair-wise comparison using DIAGNOcam and bitewing).

ELIGIBILITY:
Inclusion Criteria:

individuals who want to participate in the study ,the presence of 2 or more non-cavitated interproximal caries lesions with dark shadow involved in the enamel on the DIAGNOcam image -

Exclusion Criteria:

* patient who diagnosed with dentinogenesis imperfecta

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-12-10 (Estimated); Study Completion 2021-08-10 (Estimated)

PRIMARY OUTCOMES:
pairwise bitewing radiograph and DIAGNOcam image | after three years
  comparing the outcome of bitewing radiograph and DIAGNOcam image of pre- and post- operation

SECONDARY OUTCOMES:
compare the cost-effectiveness between resin infiltration and remineralization | after three year years
  calculate the consumption of infiltrant and Duraphat,combined with the effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: liuyan meng, dovtor, Principal Investigator — Hospital of Stomatology, Wuhan University
Locations (1):
- Wuhan university, Wuhan, Hubei, China